CLINICAL TRIAL: NCT01288651
Title: Intravenous Iron Treatment In Iron Deficient Patients With Idiopathic Pulmonary Arterial Hypertension
Brief Title: Iron Deficiency In Pulmonary Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: G. Ruiter, MD, VU university medical center, Department of Pulmonology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-247
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Iron deficiency; Exercise
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension; Iron Deficiencies; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ferricarboxymaltose — Ferricarboxymaltose (Ferinject®, Vifor Pharma) is used for intravenous iron administration. This iron is administered in high dose iron infusion of 1000 mg iron (equals 20 ml Ferinject) in 250 ml saline in the vein (infusion site)within 2 hours. During infusion, patients will be observed and blood pressure and heart rate are monitored before and after administration.
  Four weeks after iron administration, iron parameters are measured in the general practitioners setting. When iron parameters are still under normal values, a repeat infusion will be given of 500 mg iron (equals 10 ml Ferinject).

SUMMARY:
Patients with idiopathic pulmonary arterial hypertension (IPAH) and iron deficiency were previously shown to have a decreased six-minute walking distance. Therefore the investigators hypothesized that intravenous iron administration would improve exercise capacity in iron deficient IPAH patients.

30 patients will be recruited for iron infusions. At baseline and after 12 weeks (endpoint)exercise test will be performed.

DETAILED DESCRIPTION:
Background: Patients with pulmonary arterial hypertension (PAH) develop progressive right heart failure which eventually will lead to death. During progression of the disease the physical performance of the patients deteriorates. Maintaining their exercise capacity is a major goal in PAH treatment. Iron treatment is known to have a positive effect on physical performance in patients with left heart failure and iron deficiency. Whether this is also effective in patients with right heart failure (PAH) and iron deficiency is until now unknown.

Objective: To evaluate the effects of intravenous iron supplementation on exercise capacity in iron deficient IPAH patients.

Study design: Intervention study

Study population: Patients with idiopathic pulmonary arterial hypertension (IPAH) and iron deficiency

Patients receive an iron bolus infusion of 1000 mg iron after baseline measurements.

Main study parameters/endpoints:

Primary endpoint: six minute walking distance (6WMD) Secondary endpoints: cardiopulmonary exercise test, myoglobin concentration in quadriceps muscle, quadriceps muscle fiber strength, serum iron parameters, serum inflammatory parameters, quality of life (QOL), and NYHA functional class.

The patients will be hospitalised two days at the beginning and two days at the end of the study to perform the exercise and strength tests, six minute walking distance and for biopsy of the quadriceps muscle. Also NYHA functional class will be determined and a QOL questionnaire has to be filled in. After the baseline measurements an iron infusion will be given (Ferinject 1000mg).

The investigators hypothesize that iron deficient IPAH patients will benefit from iron treatment with improved exercise capacity reflected in an increased 6MWD.

ELIGIBILITY:
Inclusion Criteria:

* Stable idiopathic pulmonary arterial hypertension (stable disease for at least 3 months)
* iron deficiency (serum iron below 10 μmol/l, decreased transferrin saturation (< 15% in females and < 20% in males) and serum ferritin < 100 μg/l) irrespective of the coexistence of anaemia

Exclusion Criteria:

* Current iron therapy (oral or iv)
* Current other study medication for PAH
* History of anaemia or current treatment for anaemia
* Liver function impairment
* Chronic disease other than PAH (rheumatism, asthma, chronic infection)
* Acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
six-minute walking distance | 12 weeks
  The primary endpoint is improvement in six-minute walking distance

SECONDARY OUTCOMES:
Serum iron parameters | 0 and 12 weeks
  Serum iron parameters and inflammatory parameters are measured
Exercise capacity | 0 and 12 weeks
  Cardiopulmonary exercise testing is performed to measure maximal exercise capacity and exercise endurance time.
Quadriceps muscle function | 0 and 12 weeks
  A biopsy from the quadriceps muscle is taken for histochemical analysis, myoglobin measurements and muscle fiber strength characteristics
Cardiac Function | 0 and 12 weeks
  A cardiac MRI is performed to measure cardiac function
Quality of life | 0 and 12 weeks
  Quality of life and NYHA functional class is established.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Vonk-Noordegraaf, Prof MD PhD, Principal Investigator — VU University Medical Center, Deparment of Pulmonology
Locations (1):
- VUmc, Amsterdam, Netherlands

REFERENCES:
- [Derived] Ruiter G, Manders E, Happe CM, Schalij I, Groepenhoff H, Howard LS, Wilkins MR, Bogaard HJ, Westerhof N, van der Laarse WJ, de Man FS, Vonk-Noordegraaf A. Intravenous iron therapy in patients with idiopathic pulmonary arterial hypertension and iron deficiency. Pulm Circ. 2015 Sep;5(3):466-72. doi: 10.1086/682217. PMID 26401247